CLINICAL TRIAL: NCT04366206
Title: Factors Associated With Clinical Outcomes in Patients Hospitalized for Covid-19 in GHT-93 Est
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Intercommunal Robert Ballanger (Other)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Dr. Hélène GROS, Principal Investigator, Centre Hospitalier Intercommunal Robert Ballanger
Other Study IDs: GHTRB-2020-01
Record Dates: First submitted 2020-04-19; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: COVID; SARS-CoV 2
Keywords: covid-19; SARS-Cov-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients exposed to the study variable: Depending on the studied variable (treatment or risk factor)
- Patients not exposed to the study variable: Depending on the studied variable (treatment or risk factor)

SUMMARY:
Healthcare centers treated several hundreds of patients with Covid-19 and prospectively gathered information in electronic format between March, 2020 to April, 2020. In the course of Covid-19 treatment, physicians employed several drugs, including hydroxychloroquine, azithromycin, lopinavir/ritonavir, tocilizumab, baricitinib, sarilumab, corticosteroids and systematic antibiotics (list is not exhaustive).

This cohort study aims to assess factors associated with clinical outcomes in patients hospitalized for Covid-19, by analyzing associations between treatments and outcomes.

All data are collected in electronical records during routine practice.

DETAILED DESCRIPTION:
Healthcare centers treated several hundreds of patients with Covid-19 and prospectively gathered information in electronic format between March, 2020 to April, 2020. In the course of Covid-19 treatment, physicians employed several drugs, including hydroxychloroquine, azithromycin, lopinavir/ritonavir, tocilizumab, baricitinib, sarilumab, corticosteroids and systematic antibiotics (list is not exhaustive).

This cohort study aims to assess factors associated with clinical outcomes in patients hospitalized for Covid-19.

Risk factors which will be studied include: baseline characteristics such as medical history and drugs with corresponding administration protocols.

Main outcomes include all-cause mortality, need for mechanical ventilation, for ICU transfer and all relevant biological syndromes.

All data are collected in electronical records during routine practice and additional data may be collected retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized for Covid-19
* severe pneumonia defined as pulse O2 < 96% despite > 6L/min

Exclusion Criteria:

* lack of consent
* palliative care patients
* patients in ICU
* patients transferred from ICU

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients hospitalized for Covid-19 may be eligible to join this cohort study
Sampling Method: Non-Probability Sample
Enrollment: 143 (Estimated)
Dates: Start 2020-03-14 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Composite of death and mechanical ventilation | At 14-days follow-up
  Composite of death and mechanical ventilation

SECONDARY OUTCOMES:
Need for mechanical ventilation | At 14-days follow-up
  Need for mechanical ventilation
Death | At 14-days follow-up
  All-cause mortality
Acute kidney injury | At 14-days follow-up
  As defined by AKIN
Acute respiratory distress syndrome | At 14-days follow-up
  As defined by Berlin criteria: P/F ratio below 200, with PEEP > +5 cmH20, radiologic findings compatible with ARDS and not explained by heart failure, occurring within 7 days of an acute pulmonary or non-pulmonary aggression.
Cardiac arrhythmia and conduction disorder | At 14-days follow-up
  Documented by EKG monitoring
Composite of death and mechanical ventilation | Up to 60 days after inclusion
  Composite of death and mechanical ventilation
60-days mortality | Up to 60 days after inclusion
  All cause mortality at 60 days follow-up whenever possible
60-days mechanical ventilation | Up to 60 days after inclusion
  If patient was mechanically ventilated within 60 days of inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Gros, MD, Study Director — Robert Ballanger
Locations (2):
- France (2):
  - Centre Hospitalier Intercommunal Robert Ballanger, Aulnay-sous-Bois
  - Groupe Hospitalier Pitie Salpetriere, Paris

IPD SHARING:
Plan to Share IPD: No